CLINICAL TRIAL: NCT00860002
Title: The Benefits and Limits of Laparoscopic Surgery for Uterine Fibroids
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Peng-Hui Wang, M.D., Ph.D., Associate Professor, Department of Obstetrics and Gynecology, Taipei Veterans General Hospital
Other Study IDs: VGHIRB-98-01-20A
Record Dates: First submitted 2009-03-10; First posted 2009-03-11 (Estimated); Last update posted 2010-06-08 (Estimated); Status verified 2010-06

CONDITIONS: Uterine Fibroids
Keywords: myomectomy; uterine artery occlusion; uterine vessel occlusion; fibroids; leiomyomas; Surgical technique, patient suffering and outcomes
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (17):
- 1: Ultramini laparotomy (UMLT) myomectomy (UMLT-M) versus laparoscopic myomectomy (LM)
- 2: Laparoscopically aided myomectomy (LAM) versus LM
- 3: LAM versus UMLT-M
- 4: Mini laparotomy myomectomy (ML-M) versus UMLT-M
- 5: Laparoscopic uterine artery occlusion with blockage of anastomosis between the uterine and ovarian vessels (LUVO) versus laparoscopic uterine artery occlusion without blockage of anastomosis between the uterine and ovarian vessels (LUAO)
- 6: LUVO+LAM versus LUAO+LAM
- 7: LUVO+LM versus LUAO+LM
- 8: LUVO+UMLT-M versus LUAO+UMLT-M
- 9: LUVO versus UMLT-UVO
- 10: UMLT-UVO versus UMLT-UAO
- 11: LUAO versus UMLT-UAO
- 12: UMLT-UVO+UMLT-M versus UMLT-UAO+UMLT-M
- 13: LUVO versus LM
- 14: LUVO versus LAM
- 15: LUVO versus LUAO+LM
- 16: LUVO versus LUAO+UMLT-M
- 17: LUVO versus LUAO+LAM

SUMMARY:
Uterine leiomyomas (i.e., fibroids, myomas) are the most common gynecologic tumors in women of reproductive age (1). Clearly, the majority of such lesions are asymptomatic (2). Symptoms directly attributable to these benign tumors represent the most common reason for laparotomy in non-pregnant women in the United States (3,4), and also in Taiwan (5). Whereas in decades past, hysterectomy was seen almost as a panacea for uterine leiomyomas, more recently attention has been paid to the development of pharmaceutical agents and less-invasive procedures (6). Frequently, such procedures are designed to retain the uterus (6). Of these, myomectomy may be a choice among the uterine-sparing treatments for symptomatic uterine myoma (7,8).

The surgical mode of access usually employed in myomectomy is traditional exploratory laparotomy or its modification-mini-laparotomy (MLT) (9) or ultra-mini laparotomy (UMLT) (10,11), though recently, laparoscopy (12-14) or a combination of laparoscopy and MLT (9), vaginal surgery (15), and hysteroscopic myomectomy (16-21) have represented valid alternatives. However, myomectomy alone provides varying degrees of symptom control and a high percentage of recurrence, not only for the tumors themselves, but also for the symptoms. For example, one study reported that symptom resolution varied from 84.0% to 100% depending on different items and 21 (19.4%) of 108 patients experienced a recurrence after an average interval of 16 months (range, 1.8-47.4 months) (22). Therefore, an alternative or additional therapy might be required to provide longer durable symptom control and minimize tumor recurrence. One of the strategies is laparoscopic uterine vessel occlusion (LUVO), also known as laparoscopic uterine artery occlusion (LUAO) (23,24).

The rationale for using LUVO in the management of symptomatic myomas is found in the successful experience with uterine-artery embolization (UAE), which was introduced in 1995 as an alternative technique for treating fibroids (25). Since then it has become increasingly accepted as a minimally invasive, uterine-sparing procedure, and studies have reported the relief of excessive menstrual bleeding or pressure in 80-90% of patients (26-32). LUVO provided similar relief of symptoms (89.4% with symptomatic improvement and 21.2% with complete resolution of symptoms) in 2001 in a 7- to 12-month follow-up of 87 patients after LUVO (33).

Since that time there has been rapid growth in the use of this treatment with various modifications, such as simultaneous accompaniment with myomectomy either through laparoscopy or ML, and there has been considerable research into its outcome (22,34-42). However, in our previous data, we found that a combination of LUVO and myomectomy provided definite effectiveness in symptom control for these women with symptomatic uterine myomas (98.1% to 100% symptom resolution depending on various kinds of items), minimized tumor recurrence, and rendered the vast majority of re-interventions unnecessary (22). Myomectomy can be performed by the laparoscopic approach or by ML when patients are undergoing the LUVO procedure. Before 2002, we often used ML to perform myomectomy (22). However, we have shortened the incision to less than 4 cm, creating ultramini-laparotomy (UMLT) to perform myomectomy (10,11,43).

Since many conservative therapies might provide less or more therapeutic effects on the symptom control and disease status, the aim of this prospective study tries to evaluate the therapeutic outcomes of these symptomatic uterine myomas after different kinds of therapies in the coming 5 years at Taipei Veterans General Hospital.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic;
* having a wish to retain their uterus;
* an absence of previous abdominal or pelvic surgery;
* a number of visible uterine masses (myomas) less than or equal to 5 intramural or sub-serous myomas (without peduncle);
* a maximum diameter of no more than 8 cm;
* an absence of prominent or significant pelvic adhesion on clinical evaluation; AND
* at least a 2-year thorough follow-up record available.

Exclusion Criteria:

* without pathological diagnosis of myoma if the specimen can be obtained; OR
* any violation the above-mentioned criteria.

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women between 2009 and 2014 booked for treatment who had symptomatic uterine myomas, will be included in the present study. All the treatments for symptomatic uterine myomas, including medical treatment with different kinds of medication, and uterine-sparing surgery including myomectomy, which is performed through traditional exploratory laparotomy (LT), mini-laparotomy (MLT), ultramini-laparotomy (UMLT), laparoscopy (L), the vagina (V) or hysteroscopy (H), and LUVO and combination therapy, and the definite treatment of hysterectomy, through different routes, such as vagina, laparoscopic assistance, and convention exploratory laparotomy. All patients should have uterine fibroids with symptoms, comprising either menstrual problems such as menorrhagia and pain, or compression syndrome, including a bulge-like sensation and frequency. These women will be informed that they can choose to be treated with any one of the above-mentioned procedures, based on their willingness and preference.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Surgical technique, patient suffering, and outcomes (symptom control, relapse of symptoms, re-intervention, regularity of menstrual cycles and pregnancy outcome) in both groups. | 2-years and 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Peng-Hui Wang, 201, Section 2, Shih-Pai Road, Taipei, Taipei, Taiwan